CLINICAL TRIAL: NCT01200732
Title: Clinical Efficacy of Phosphodiesterase-5 Inhibitor Tadalafil in Eisenmenger Syndrome - A Randomised, Placebo Controlled, Double Blind, Crossover Study
Brief Title: Phosphodiesterase-5 Inhibitor in Eisenmenger Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: saibal mukhopadhyay, Govind Ballabh Pant Hospital,Delhi university
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ES/F.501(134)/EC/07/MC
Record Dates: First submitted 2010-09-08; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-08

CONDITIONS: Eisenmenger Syndrome
Keywords: Tadalafil; phosphodiesterase-5 inhibitor; Eisenmenger syndrome
MeSH Terms: conditions — Eisenmenger Complex | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Active Comparator)
  Interventions: Drug: Tadalafil, placebo
- placebo (Placebo Comparator)
  Interventions: Drug: Tadalafil, placebo

INTERVENTIONS:
Drug: Tadalafil, placebo — 20mg tablets, 2 tablets Once daily(i.e 40mg once daily) 20mg placebo 2 tablets once daily

SUMMARY:
A preliminary observational study by the investigators has shown that tadalafil, a selective phosphodiesterase-5 inhibitor (PDE-5) decreases pulmonary vascular resistance(PVR) in patients of eisenmenger syndrome (ES) resulting in increase in pulmonary blood flow (Qp), systemic oxygen saturation (SaO2), functional class and exercise capacity. The aim of this placebo controlled trial was to assess the effect of the drug on exercise capacity and functional class compared to placebo.

DETAILED DESCRIPTION:
Methods Patients of ES with age greater than or equal to 18 years and weight greater than or equal to 30 kgs in World Health Organisation (WHO) functional class II and III attending our congenital clinic were invited to participate in the study. Informed written consent was taken from all the patients before screening procedures were initiated for the study. A detailed clinical examination and non-invasive testing including electrocardiogram, chest X ray, pulmonary function tests (to exclude associated restrictive/obstructive lung disease) and echocardiography(including contrast echo if required for demonstrating right to left shunt) were conducted. Patients with simple congenital heart defects (atrial septal defect > 2cm, ventricular septal defect > 1cm and aortopulmonary communications > 0.4 cm) with echocardiographic evidence of right to left shunt were included. Medical therapy and clinical condition of the patients had to be stable for 3 months prior to screening. Patients on treatment with prostanoids, endothelial receptor antagonists (ERA), PDE-5 inhibitors or any other vasodilators with in 1month prior to screening were excluded. A systemic pulse oximetry (SpO2) between 70% and 90% at rest in room air and a baseline 6 minute walk test(6MWT) distance between 150 and 450 meters were required for inclusion. Eisenmenger physiology was confirmed by cardiac catheterization as mean pulmonary artery pressure > 40mmHg, pulmonary capillary wedge pressure < 15mmHg and pulmonary vascular resistance >10 wood units/m2. Oxygen study was also done in selected patients to diagnose reversible pulmonary arterial hypertension(PAH) and such patients were excluded. Patients were also excluded if they were in WHO class IV, were in congestive heart failure or had PCWP > 15mmHg,had left ventricular ejection fraction <40%, atrial fibrillation, patent ductus arteriosus, complex congenital heart defects, restrictive lung disease(total lung capacity < 70% of predicted), obstructive lung disease ( forced expiratory volume in 1 second [FEV1] < 70% of predicted with FEV1/ Forced vital capacity [FVC] < 60%), previously diagnosed coronary artery disease requiring nitrate therapy, abnormal biochemical profile and hypersensitivity to PDE- 5 inhibitors. Left and right heart catheterization was done in eligible patients as described in our preliminary observational study. Calculation of pulmonary and systemic blood flow(Qs), PVR and SVR was performed using the Ficks equation and assumed values of oxygen consumption according to age and gender of patient. The study was conducted according to the most recent amendments to the Declaration of Helsinki and in adherence to good clinical practice guidelines. The trial was approved by the National Drug Regulatory Authority (DCG) and the ethical committee of our institution.

Study design and procedure:

A double blind randomised placebo controlled crossover trial was carried out to study the efficacy and safety of oral tadalafil. Eligible patients were randomised to receive either oral tadalafil or matching placebo after baseline assessment of WHO functional class, exercise capacity by 6MWT and hemodynamic study by cardiac catheterization. Randomisation, blinding and drug/placebo administration was done by two pharmacists of the hospital. Patients received tadalafil 40mg once daily or matching placebo for 6 weeks which was followed by a 2 week washout before crossing over to the other drug for another 6 weeks. Routine medications for PAH like digoxin and diuretics was continued through out the study. Compliance was assessed by the pill count method at 3 weekly intervals. Safety of the drug or placebo was assessed by noting adverse effects, vital signs and (SaO2) by pulse oximetry at 3 week intervals. Clinical assessments (WHO functional class), 6 MWT and hemodynamic parameters by cardiac catheterization were reassessed after 6 weeks and again at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ES with age greater than or equal to 14 years and weight greater than or equal to 30 kgs in World Health Organisation (WHO) functional class II and III attending our congenital clinic were invited to participate in the study

Exclusion Criteria:

* WHO class IV,
* congestive heart failure or had PCWP > 15mmHg,
* left ventricular ejection fraction <40%,
* atrial fibrillation,
* patent ductus arteriosus,
* complex congenital heart defects,
* restrictive lung disease(total lung capacity < 70% of predicted), obstructive lung disease ( forced expiratory volume in 1 second [FEV1] < 70% of predicted with FEV1/ Forced vital capacity [FVC] < 60%),
* previously diagnosed coronary artery disease requiring nitrate therapy,
* abnormal biochemical profile and
* hypersensitivity to PDE- 5 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The primary end point of efficacy was improvement in exercise tolerance as assessed by the un-encouraged 6 minute walk test (6MWT) compared to baseline after 6 weeks of treatment | 6 weeks

SECONDARY OUTCOMES:
The secondary endpoints were effect of the drug on systemic oxygen saturation (SaO2) | 6 weeks
The secondary endpoints were effect of the drug on effective pulmonary blood flow(EPBF) | 6 weeks
The secondary endpoints were effect of the drug on pulmonary vascular resistance (PVR). | 6 weeks
The secondary endpoints were effect of the drug on systemic vascular resistance (SVR) | 6 weeks
The secondary endpoints were effect of the drug on WHO functional class | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Saibal Mukhopadhyay, M.D;D.M, Principal Investigator — GBPant Hospital; Sanjay Tyagi, M.D;D.M, Study Director — GBPant Hospital
Locations (1):
- Govind Ballabh Pant Hospital(GB Pant Hospital), New Delhi, New Delhi, India

REFERENCES:
- [Background] Mukhopadhyay S, Sharma M, Ramakrishnan S, Yusuf J, Gupta MD, Bhamri N, Trehan V, Tyagi S. Phosphodiesterase-5 inhibitor in Eisenmenger syndrome: a preliminary observational study. Circulation. 2006 Oct 24;114(17):1807-10. doi: 10.1161/CIRCULATIONAHA.105.603001. Epub 2006 Oct 9. PMID 17030688
- [Derived] Mukhopadhyay S, Nathani S, Yusuf J, Shrimal D, Tyagi S. Clinical efficacy of phosphodiesterase-5 inhibitor tadalafil in Eisenmenger syndrome--a randomized, placebo-controlled, double-blind crossover study. Congenit Heart Dis. 2011 Sep-Oct;6(5):424-31. doi: 10.1111/j.1747-0803.2011.00561.x. PMID 21914136